CLINICAL TRIAL: NCT07280572
Title: RECLAIM: an Adaptive Platform Trial for the Evaluation of Treatments for Post-Acute Sequelae of SARS-CoV-2 Infection (PASC)
Brief Title: RECLAIM Adaptive Platform Trial for PCC Treatments
Acronym: RECLAIM
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Janneke van de Wijgert (Other)
Collaborators: European Clinical Research Alliance for Infectious Diseases (ECRAID) (Other)
Responsible Party: Sponsor-Investigator, Janneke van de Wijgert, Professor, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUCT 2024-511580-28; D-25-500086 (Other: NedMec Medical Research Ethics Committee, Utrecht, Netherlands)
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Post COVID Condition
Keywords: Post COVID condition; Clinical trial; Intervention; Repurposed drugs; Metformin; Colchicine; PAIS; Post Acute Sequelae of COVID-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Metformin; Colchicine

STUDY DESIGN:
Masking Description: The first domain is open label. The second domain (minocyclin versus placebo) will be placebo-controlled and blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Usual care (No Intervention): Participants receive their standard of care for PCC, without starting any new medications during study participation.
- Metformin (Experimental)
  Interventions: Drug: Metformin
- Colchicine (Experimental)
  Interventions: Drug: colchicine

INTERVENTIONS:
Drug: Metformin — Participants receive metformin tablets for a period of 12-weeks.
  Arms: Metformin
Drug: colchicine — Participants receive colchicine tablets for a period of 12-weeks.
  Arms: Colchicine

SUMMARY:
RECLAIM is a Phase III, multi-domain, randomized, controlled, adaptive platform trial, designed to evaluate efficacy and safety of repurposed medications in patients with post-COVID condition (PCC). The trial started in the Netherlands in February 2025, comparing metformin, colchicine and usual care in an open-label domain. The information in this registration concerns that first domain in the Netherlands. A second domain, comparing minocyclin to a matching placebo, is expected to start in January 2026, also in the Netherlands. Trial-arms, additional domains and implementing countries may be introduced or terminated as the trial progresses. Participation is fully remote, using electronic consenting, video consultations and home delivery of medication. Default IP use is 12 weeks with biweekly online follow-up questionnaires between Day-1 and Week-12, and one final follow-up questionnaire at week-24.

ELIGIBILITY:
Inclusion criteria

1. Adults aged 18 years or older.
2. Residing in the Netherlands (but excluding the Carribbean parts of the Netherlands) for the duration of trial participation.
3. Persistent PCC symptoms, including fatigue and/or PEM, for a period of at least 12 weeks after the onset of a SARS-CoV-2 infection. The symptoms were not present prior to the infection, but may have partially subsided and resurged after the infection.
4. Self-reported confirmation of having had a SARS-CoV-2 infection by:

   1. Positive SARS-CoV-2 nucleic acid amplification test, such as PCR;
   2. Positive SARS-CoV-2 rapid diagnostic test, including home-administered tests;
   3. COVID-19 diagnosis by a medical specialist (GP or in-hospital), based on the above or other clinical tests and assessments.

   The above information will not be verified in medical records.
5. Willing and able to provide informed consent.
6. Willing and able to perform trial procedures.
7. Allowing their GP/treating physicians/pharmacy and the RECLAIM trial team to exchange medical information that is relevant for the participant's safety and trial assessments.

Exclusion criteria:

1. Having been diagnosed with (exacerbation of) a chronic disease that can account for the onset of the PCC-like symptoms.
2. Being hospitalized or institutionalized at screening. Patients can be rescreened after discharge.
3. Presence of a serious medical condition that would prevent completion of follow-up.
4. Currently enrolled, or having been enrolled within the last 30 days, in any other study where that study's interventions or procedures may affect RECLAIM outcomes or procedures. Individuals can be rescreened after at least 30 days have passed since participation in such a study has been completed.

   The following exclusion criteria will apply to all potential participants WITHIN ONE TRIAL DOMAIN (these patients may still qualify for another trial domain):
5. The participant cannot be randomized to at least one IP arm and its control arm within a trial domain due to:

   1. Known hypersensitivity to an active IP ingredient or IP/placebo excipient;
   2. Receiving a treatment that is contraindicated to a trial IP;
   3. Already using a trial IP, or a drug in the same drug class as a trial IP, outside of the trial;
   4. Any other reason why a trial IP cannot be used, such as (risk of) pregnancy or breastfeeding or renal insufficiency.

During screening, these criteria will be assessed by licensed trial physicians. They will question the patient and verify prescription drug and contraceptive use, and other medical exclusion criteria, in each individual patient's medical and/or pharmacy records. The absence of pregnancy in women of childbearing potential has to be confirmed by a negative urine or serum pregnancy test.

Additional IP-specific in- and exclusion criteria, if any, are listed in relevant treatment-specific appendices to the core protocol. These also describe the latest information about drug interactions and contraindications as per the IP's SmPC/PIL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Physical health-related quality of life (HRQoL) | 12 weeks
  PROMIS-29 physical health summary score

SECONDARY OUTCOMES:
Mental HRQoL | 12 weeks
  PROMIS-29 mental health summary score
Other aspects of HRQoL | 12 weeks
  PROMIS-29 domain scores: physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, sleep disturbance.
Fatigue | 12 weeks
  Checklist Individual Strength, fatigue severity subscale (CIS-8)
Post Exertional Malaise (PEM) | 12 weeks
  DePaul Symptom Questionnaire (DSQ-2) PEM questions
Cognitive functioning | 12 weeks
  PROMIS cognitive function 8a
Post Orthostatic Tachycardia Syndrome (POTS) | 12 weeks
  DSQ-2 POTS questions
Safety of IPs | 12 weeks
  Frequency of related and unrelated (S)AEs and SUSARs in each IP arm including their severity and outcome.
Tolerability of IPs | 12 weeks
  Level of adherence to each IP. Percent of participants with adequate adherence for the specific IP.
Durability of IP treatment responses | 24 weeks
  The proportion of participants that maintain HRQoL treatment success at 24 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Julius Center for Health Sciences and Primary Care University Medical Center Utrecht, Netherlands, Utrecht, Netherlands